CLINICAL TRIAL: NCT04852757
Title: Estimating the Prevalence of Postpartum Anxiety and Depression in the Context of the COVID-19 Pandemic
Brief Title: Estimating the Prevalence of Postpartum Anxiety and Depression in the Context of the Coronavirus Disease (COVID-19) Pandemic
Acronym: PsyCOVIDUM
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PsyCOVIDUM
Record Dates: First submitted 2021-04-20; First posted 2021-04-21 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Depression, Postpartum
Keywords: Covid19
MeSH Terms: conditions — Depression, Postpartum; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In December 2019, infection with a new coronavirus Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) emerged in China and has since spread throughout the world. Forms of varying severity of COVID-19, a disease induced by this emerging virus, have been described in pregnant women. In addition to the direct effects of the virus on the pregnant woman and the fetus, the pandemic context itself is likely to act as a psychological risk factor and to alter the protective factors for mental disorders. This pandemic context is in itself anxiety-provoking, even traumatogenic, particularly because of the potentially lethal infectious risk that it conveys, all the more so in psychologically vulnerable populations. In addition to the fear of viral contamination, the fear of childbirth and the postpartum period, which includes a more or less important part of anxiety-provoking uncertainty, is added to the fear of viral contamination in the perinatal period. This addition of stress factors is likely to increase the prevalence of perinatal depressive disorders and anxiety disorders, particularly the psychotraumatic experience of childbirth. Sanitary and social measures, such as quarantine, restriction of access of accompanying persons to maternity unit, or contagious isolation of mothers suspected of being infected or infected, which may furthermore impose a separation of mother and child, are also likely to have psychopathological consequences.

In this context, three maternity wards of the PREMA University Hospital Federation (UHF PREMA) : Groupe hospitalier Paris Saint-Joseph (GHPSJ), Louis Mourier Hospital (APHP) and Port-Royal Hospital (APHP), in partnership with the "Centre de Psychopathologie du Boulevard Brune (CPBB)" and the psychiatry department of the Louis Mourier Hospital have set up a care protocol consisting of a systematic screening offered to women following childbirth on the first day of their pregnancy, aimed at identifying those with perinatal anxiety and depressive symptoms. Women presenting symptoms are then treated according to the modalities adapted to the organization of each of these three centers.

DETAILED DESCRIPTION:
Screening in these three centers is based on the use of a self-administered questionnaire for the detection of depressive disorders, the Edinburgh Postnatal Depression Scale (EPDS), which allows the calculation of a score.

In addition to the EPDS, three other tools are used at the GHPSJ maternity : a questionnaire to screen for anxiety, the State-Trait Anxiety Inventory (STAI-S), and two for trauma symptoms, the Peritraumatic Dissociative Experiences Questionnaire (PDEQ) and the Peritraumatic Distress Inventory (PDI). In this center, the screening includes a second phase with a home mailing between 6 and 8 weeks after delivery: the EPDS, the STAI-S and the Impact Events Scale-Revised (IES-R), another test screening for post-traumatic stress.

Based on the protocol implemented in these three maternity hospitals, the present research project aims to estimate the prevalence of postpartum depressive disorders at different times during and after the COVID-19 pandemic. It will also aim to identify the factors associated with the occurrence of these disorders, primarily to determine the association between elements of the pandemic context and the risk of postpartum depressive and anxiety disorders.

This project, which is based on an epidemiological approach, thus aims to assess the mental health risks associated with the COVID-19 pandemic. Postpartum women are a particularly vulnerable group, especially in terms of mental health.

Indeed, 1 to 5% develop post-traumatic stress disorder during this period and 10 to 20% develop post-partum depression. Furthermore, the National Confidential Survey on Maternal Deaths (NCSMD) shows that suicide is now the leading cause of maternal death in France (i.e., death occurring between conception and the first year following birth), before postpartum hemorrhage and before preeclampsia (data not yet published). From pooled English, Dutch, and French data, we observe that 36% of maternal deaths occurring between conception and the first year postpartum are deaths by suicide.

The COVID-19 pandemic and the associated measures that went as far as confining the population were very likely to increase the factors favouring the occurrence of mental health impairment in the general population, but perhaps even more so in certain at-risk groups such as postpartum women.

The pandemic context, whether through the fears associated with the viral infection for oneself or one's family, or through the consequences of the exceptional measures put in place in many countries to limit viral circulation, has had an effect on the general population and on the population of women in pregnancy, in different contexts. To date and to our knowledge, there is no data that would allow us to know the impact that this context may have had on the mental health of pregnant women in France. Moreover, there are no studies, either in France or elsewhere, on the impact of this pandemic context on the prevalence of psychological disorders in the postpartum period. However, this period is already a time of particular psychological vulnerability, a time when the risk of maternal suicide is at its highest. It is moreover reasonable to think that the pandemic impact and the general and local measures that accompany it may have an even greater impact during this postpartum period. The measures taken to prevent and protect against viral dissemination have had the effect of completely closing most maternity services to fathers and thus depriving mothers, totally or partially, of social and marital support and, in some situations, of physical proximity to their children, all of which are risk factors for postpartum depression.

In the perinatal context, it has also been documented that post-traumatic stress disorder is strongly associated with the risk of perinatal depression.

ELIGIBILITY:
Inclusion Criteria:

* Adult pregnant women delivering after 24 weeks of amenorrhea between April 6, 2020 and the end of the COVID-19 epidemic in one of the three participating maternity units
* French speaking patient

Exclusion Criteria:

* Situation of fetal death or Medical Interruption of Pregnancy
* Patient under guardianship or curators
* Patient deprived of liberty
* Patient under court protection
* Patient opposing the use of his data for this research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult pregnant women delivering after 24 weeks of amenorrhea between April 6, 2020 and the end of the COVID-19 epidemic in one of the three participating maternity units
Sampling Method: Non-Probability Sample
Enrollment: 2580 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Follow the evolution of the prevalence of women in immediate postpartum presenting a depressive and/or anxious symptomatology in the population of 3 maternity units in the Paris area | 2 months
  Evolution during pandemic fluctuations of the proportion of women with a positive screen for anxiety and/or depressive disorders in the immediate postpartum

SECONDARY OUTCOMES:
Estimate the prevalence, in the context of a COVID-19 pandemic, of women in the immediate postpartum period presenting depressive and/or anxious symptoms (EPDS) in the population of women giving birth (in the 3 hospitals) | Day 3
  Prevalence of women with immediate postpartum EPDS >10.
Estimate, in the context of a COVID-19 pandemic, the prevalence of women in the immediate postpartum period presenting depressive and/or anxious symptoms (STAI-S) in the population of women giving birth (in the 3 hospitals) | Day 3
  Prevalence of women with immediate postpartum (STAI-S) > 45
Estimate, in the context of a COVID-19 pandemic, the prevalence of women in the immediate postpartum period presenting depressive and/or anxious symptoms (PDEQ) in the population of women giving birth (in the 3 hospitals) | Day 3
  Prevalence of women with immediate postpartum Peritraumatic Dissociative Experiences Questionnaire (PDEQ) > 15
Estimate, in the context of a COVID-19 pandemic, the prevalence of women in the immediate postpartum period presenting depressive and/or anxious symptoms (PDI) in the population of women giving birth (in the 3 hospitals) | Day 3
  Prevalence of women with immediate postpartum Peritraumatic Distress Inventory scale (PDI) > 15
Estimate in the context of a COVID-19 pandemic the prevalence of women at 2 months postpartum with depressive and/or anxious symptoms (EPDS) in the population of women giving birth at the GhPSJ maternity hospital | 2 months
  Prevalence of women with immediate postpartum EPDS >10
Estimate in the context of a COVID-19 pandemic the prevalence of women at 2 months postpartum with depressive and/or anxious symptoms (STAI-S) in the population of women giving birth at the GhPSJ maternity hospital | 2 months
  Prevalence of women with immediate postpartum (STAI-S) > 45
Estimate in the context of a COVID-19 pandemic the prevalence of women at 2 months postpartum with depressive and/or anxious symptoms (PDEQ) in the population of women giving birth at the GhPSJ maternity hospital | 2 months
  Prevalence of women with immediate postpartum Peritraumatic Dissociative Experiences Questionnaire (PDEQ) > 15
Estimate in the context of a COVID-19 pandemic the prevalence of women at 2 months postpartum with depressive and/or anxious symptoms (IES-R) in the population of women giving birth at the GhPSJ maternity hospital | 2 months
  Prevalence of women with immediate postpartum Impact Events Scale-Revised (IES-R) > 12
Investigate factors associated with the risk of developing depressive and/or anxiety symptomatology in the COVID-19 pandemic context | 3 days to 2 months
  Measure of association between COVID-19 infection and risk of having a score above the cutoff
Investigate factors associated with the risk of developing depressive and/or anxiety symptomatology in the COVID-19 pandemic context | 3 days to 2 months
  Measure of association between time of delivery (reflecting exposure to general and local quarantine, as well as risk of viral infection) and risk of having a score above the cutoff
Investigate factors associated with the risk of developing depressive and/or anxiety symptomatology in the COVID-19 pandemic context | 3 days to 2 months
  Measure of association between maternal socio-familial isolation in the postpartum period and the risk of having a score above the cutoff
Investigate factors associated with the risk of developing depressive and/or anxiety symptomatology in the COVID-19 pandemic context | 3 days to 2 months
  Measure of association between mother-child separation in the postpartum period and risk of having a score above the cutoff
Comparison of the prevalence of anxiety and depressive disorders among women not infected with SARS-CoV2 in PsyCOVIDUM with those infected in the COROPREG study (COVID-19 and pregnancy: a population-based cohort of women and newborns) | 2 months
  Measuring the impact of maternal COVID-19 infection on anxiety-depressive symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Elie AZRIA, Pr, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France